CLINICAL TRIAL: NCT02385071
Title: A Phase 1, Open-label, Randomized, 2-panel, 3-way Crossover Study in Healthy Adult Subjects to Assess the Relative Bioavailability of Simeprevir Following Single Dose Administration of Age-appropriate Oral Formulation Candidates, Compared to the 150-mg Oral Capsule, and to Assess the Effect of Food on the Bioavailability of Simeprevir Following Single Dose Administration of a Selected Age-appropriate Oral Formulation Candidate
Brief Title: A Crossover Study to Evaluate Relative Bioavailability of Simeprevir Age-appropriate Oral Formulation Candidates Compared With 150-milligram (mg) Oral Capsule in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR106516; TMC435HPC1010 (Other: Janssen Sciences Ireland UC); 2014-005448-17 (EudraCT Number)
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Healthy; Simeprevir; Bioavailability
MeSH Terms: interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (12):
- Panel1: Sequence 1 (ABC) (Experimental): Participants will receive Treatment A (150 milligram (mg) simeprevir (SMV) capsule with water under fed conditions) in Period 1; followed by Treatment B (3*50 mg capsules of SMV [including 50 mini-tablets of 1 mg each] with water under fed conditions) in Period 2; followed by Treatment C (3*50 mg dispersible SMV tablets dispersed in water under fed conditions) in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel1: Sequence 2 (BCA) (Experimental): Participants will receive Treatment B in Period 1; followed by Treatment C in Period 2; followed by Treatment A in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel1: Sequence 3 (CAB) (Experimental): Participants will receive Treatment C in Period 1; followed by Treatment A in Period 2; followed by Treatment B in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel1: Sequence 4 (CBA) (Experimental): Participants will receive Treatment C in Period 1; followed by Treatment B in Period 2; followed by Treatment A in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel1: Sequence 5 (BAC) (Experimental): Participants will receive Treatment B in Period 1; followed by Treatment A in Period 2; followed by Treatment C in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel1: Sequence 6 (ACB) (Experimental): Participants will receive Treatment A in Period 1; followed by Treatment C in Period 2; followed by Treatment B in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Panel 2: Sequence 1 (DEF) (Experimental): Participants will receive Treatment D (3*50 mg SMV capsules [including 50 mini-tablets of 1 mg each] with water or 3*50 mg dispersible SMV tablets dispersed in water under fed conditions) in Period 1; followed by Treatment E (3*50 mg SMV capsules [including 50 mini-tablets of 1 mg each] with water or 3*50 mg dispersible SMV tablets dispersed in water under fasted conditions) in Period 2; followed by Treatment F (3*50 mg SMV capsules [including 50 mini-tablets of 1 mg each] with yoghurt or 3*50 mg dispersible SMV tablets dispersed in apple juice under fed conditions) in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel 2: Sequence 2 (EFD) (Experimental): Participants will receive Treatment E in Period 1; followed by Treatment F in Period 2; followed by Treatment D in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel 2: Sequence 3 (FDE) (Experimental): Participants will receive Treatment F in Period 1; followed by Treatment D in Period 2; followed by Treatment E in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel 2: Sequence 4 (FED) (Experimental): Participants will receive Treatment F in Period 1; followed by Treatment E in Period 2; followed by Treatment D in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel 2: Sequence 5 (EDF) (Experimental): Participants will receive Treatment E in Period 1; followed by Treatment D in Period 2; followed by Treatment F in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Panel 2: Sequence 6 (DFE) (Experimental): Participants will receive Treatment D in Period 1; followed by Treatment F in Period 2; followed by Treatment E in Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F

INTERVENTIONS:
Drug: Treatment A — 150 milligram (mg) SMV capsule with water under fed conditions.
  Other Names: simeprevir
  Arms: Panel1: Sequence 1 (ABC); Panel1: Sequence 2 (BCA); Panel1: Sequence 3 (CAB); Panel1: Sequence 4 (CBA); Panel1: Sequence 5 (BAC); Panel1: Sequence 6 (ACB)
Drug: Treatment B — Treatment B (3*50 mg capsules of SMV (including 50 mini-tablets of 1 mg each) with water under fed conditions.
  Other Names: simeprevir
  Arms: Panel1: Sequence 1 (ABC); Panel1: Sequence 2 (BCA); Panel1: Sequence 3 (CAB); Panel1: Sequence 4 (CBA); Panel1: Sequence 5 (BAC); Panel1: Sequence 6 (ACB)
Drug: Treatment C — Treatment C (3*50 mg dispersible SMV tablets dispersed in water under fed conditions).
  Other Names: simeprevir
  Arms: Panel1: Sequence 1 (ABC); Panel1: Sequence 2 (BCA); Panel1: Sequence 3 (CAB); Panel1: Sequence 4 (CBA); Panel1: Sequence 5 (BAC); Panel1: Sequence 6 (ACB)
Drug: Treatment D — *50 mg SMV capsules (including 50 mini-tablets of 1 mg each) with water or 3*50 mg dispersible SMV tablets dispersed in water under fed conditions.
  Other Names: simeprevir
  Arms: Panel 2: Sequence 1 (DEF); Panel 2: Sequence 2 (EFD); Panel 2: Sequence 3 (FDE); Panel 2: Sequence 4 (FED); Panel 2: Sequence 5 (EDF); Panel 2: Sequence 6 (DFE)
Drug: Treatment E — 3*50 mg SMV capsules (including 50 mini-tablets of 1 mg each) with water or 3*50 mg dispersible SMV tablets dispersed in water under fasted conditions.
  Other Names: simeprevir
  Arms: Panel 2: Sequence 1 (DEF); Panel 2: Sequence 2 (EFD); Panel 2: Sequence 3 (FDE); Panel 2: Sequence 4 (FED); Panel 2: Sequence 5 (EDF); Panel 2: Sequence 6 (DFE)
Drug: Treatment F — 3*50 mg SMV capsules (including 50 mini-tablets of 1 mg each) with yoghurt or 3*50 mg dispersible SMV tablets dispersed in apple juice under fed conditions.
  Other Names: simeprevir
  Arms: Panel 2: Sequence 1 (DEF); Panel 2: Sequence 2 (EFD); Panel 2: Sequence 3 (FDE); Panel 2: Sequence 4 (FED); Panel 2: Sequence 5 (EDF); Panel 2: Sequence 6 (DFE)

SUMMARY:
The purpose of this study is to assess the relative bioavailability (the extent to which a drug or other substance becomes available to the body) of simeprevir (SMV) following single dose administration of age-appropriate oral formulation candidates compared to the 150 milligram (mg) capsule, and to assess the effect of food on the bioavailability of SMV following single dose administration of a selected age-appropriate oral formulation candidate.

DETAILED DESCRIPTION:
This is a Phase 1, open-label (all people know the identity of the intervention), randomized (study medication assigned to participants by chance), 2-panel, 3-way crossover (participants will receive different interventions sequentially during the trial) study in healthy adult participants. Participants will be equally divided over 2 panels, and will not be randomized between panels. Participants will not be allowed to switch panels. The study consists of 3 parts: Screening Phase (that is, 28 days before study commences on Day 1); Open-label Treatment (in subsequent 3-treatment periods in each Panel, each separated with washout period of 7 days); and Post-Treatment Phase (up to 7 days after last study drug intake). The duration of the study per participant will be at least 19 days, screening and follow-up not included. All the eligible participants will be randomly assigned to 1 of the 6 treatment sequences in each Panel. In fasted conditions, study drug will be administered following a 10-hour overnight fast. In fed conditions, participants will also fast from food for 10 hours, but will consume a high fat/high calorie breakfast within a 30-minute period. Study drug will be administered 30 minutes after the start of breakfast. Participants will not be allowed to have food until at least 4 hours after study drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Relative bioavailability of SMV formulations will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy on the basis of physical examination, medical history, 12-lead electrocardiogram (ECG) and vital signs performed at screening (after signing the ICF), and on Day -1 of the first treatment session, if applicable. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents
* Participants must be willing and able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Female participants, except for postmenopausal women, should have a negative serum pregnancy test at screening
* All female participants should have a negative urine pregnancy test on Day -1 of the first treatment session
* Male participants heterosexually active with a woman of childbearing potential must agree to use two effective methods of birth control and all men must not donate sperm during the study and for at least 30 days after receiving the last dose of study drug

Exclusion Criteria:

* Female participants who are pregnant or breast feeding at screening or on Day -1 of the first treatment session
* Participants with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin [IgM]), or hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C infection (confirmed by HCV antibody), or human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection
* Participants with a history or evidence of current or past abuse of alcohol, or recreational or narcotic drugs, which in the Investigator's opinion would compromise the participant's safety and/or compliance with the study procedures
* Participants with any history of clinically relevant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Participants with known allergies, hypersensitivity, or intolerance to simeprevir (SMV) or any of the excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Simeprevir (SMV) | Baseline up to 72 hours post-administration of study drug
  The Cmax is the maximum observed plasma concentration of SMV.
Time to Reach the Maximum Plasma Concentration (Tmax) of SMV | Baseline up to 72 hours post-administration of study drug
  The Tmax is the time to reach the maximum observed plasma concentration of SMV.
Area Under the Plasma Concentration-Time Curve From 0 to last (AUC[0-last]) Post Dose of SMV | Baseline up to 72 hours post-administration of study drug
  AUC (0-last) from time 0 to the time of the last measurable (non-below quantification limit [BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of SMV | Baseline up to 72 hours post-administration of study drug
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda [z]) of SMV | Baseline up to 72 hours post-administration of study drug
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Terminal Half-life (t[1/2]) of SMV | Baseline up to 72 hours post-administration of study drug
  The t(1/2) is defined as 0.693/Lambda (z).

SECONDARY OUTCOMES:
Number of Participants within Each Category of Taste Questionnaire | 5 to 15 minutes post administration of study drug (up to Day 19)
  Participants will assess the palatability of the SMV formulations by Taste Questionnaire, Question 1 will assess sweetness, bitterness, flavor and overall taste of the formulation; and Question 2 consists of visual analog scale wherein participants will put a cross in the box beneath the scores, corresponding to the 5-point hedonic scale (dislike it very much; dislike it a little; not sure, like it a little, like it very much).
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (7 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Harrow, United Kingdom